CLINICAL TRIAL: NCT07040670
Title: Comparison of the Diagnostic Yield and Safety Between Confocal Laser Endomicroscopy-Assisted Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration and Endobronchial Ultrasound-Guided Transbronchial Mediastinal Cryobiopsy: a Randomised Controlled Trial
Brief Title: Diagnostic Yield and Safety of Confocal Laser Endomicroscopy-Assisted Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration
Acronym: COLLEBERATIONⅢ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Deputy Director of the Department of Pulmonary and Critical Care Medicine, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2025-COLLEBERATION-Ⅲ
Record Dates: First submitted 2025-06-08; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Mediastinal Lymphadenopathies
Keywords: EBUS-TBNA; Confocal laser endomicroscopy; EBUS-TBMC

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CLE-assisted EBUS-TBNA (Experimental): Patients in this arm receive CLE-assisted EBUS-TBNA
  Interventions: Procedure: Confocal laser endomicroscopy-assisted endobronchial ultrasound-guided transbronchial needle aspiration
- EBUS-TBMC (Placebo Comparator): Patients in this arm receive EBUS-TBMC
  Interventions: Procedure: Endobronchial ultrsound-guided Mediastinal cryobiopsy

INTERVENTIONS:
Procedure: Confocal laser endomicroscopy-assisted endobronchial ultrasound-guided transbronchial needle aspiration — First, use the EBUS needle to create a hole in the airway wall. Then, insert the CLE into the lymph node via this hole and detect the lymph node. When the specific pathological finding is detected by CLE, record the location. Finally, using the needle to perform EBUS-TBNA in the area under EBUS guidance.
  Arms: CLE-assisted EBUS-TBNA
Procedure: Endobronchial ultrsound-guided Mediastinal cryobiopsy — Using the cryoprobe to perform EBUS-TBMC three times per person.
  Arms: EBUS-TBMC

SUMMARY:
Comparison of the Diagnostic Yield and Safety Between Confocal Laser Endomicroscopy-Assisted Endobronchial Ultrasound-Guided Transbronchial Needle Aspiration and Endobronchial Ultrasound-Guided Transbronchial Mediastinal Cryobiopsy in patients with mediastinal and/or hilar lymphadenopathy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old
2. Patients with at least one mediastinal and/or hilar lymphadenopathy (≥1cm in the short axis) without a known or suspected primary lung cancer, required diagnostic bronchoscopy
3. The selected patients should complete the routine examination of EBUS-TBNA/EBUS-TBMC via a tunnel before operation, such as blood routine examination, coagulation function, electrocardiogram, chest CT, etc
4. There was no contraindication of puncture and cryobiopsy
5. Fully informed of the purpose and method of the study, agreed to participate in the study, and signed the informed consent form.

Exclusion Criteria:

1. The lesion is a mediastinal cyst or abscess
2. The patient is allergic to lidocaine and midazolam （3) The site to be biopsied has a high risk of bleeding detected by Doppler and/or contrast CT such as bronchial artery penetration or suspected lung metastasis of renal cancer (4) Unstable angina pectoris, congestive heart failure, severe bronchial asthma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | On day 7 after procedure to obtain the pathological findings.
  The proportion of all individuals undergoing the diagnostic procedure under evaluation in whom a specific diagnosis is established based on the consensus definition.